CLINICAL TRIAL: NCT04991870
Title: A Phase I Clinical Trial With a Window-of-Opportunity Component of Engineered NK Cells Containing Deleted TGF-ßR2 and NR3C1 in Recurrent Grade 4 Astrocytoma (Glioblastoma)
Brief Title: Phase I CB-NK-TGF-ßR2-/NR3C1- in rGBM
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 2020-0960; NCI-2021-00598 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2020-0960 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2021-02-24; First posted 2021-08-05 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Recurrent Gliosarcoma; Recurrent Supratentorial Glioblastoma; Supratentorial Gliosarcoma
MeSH Terms: conditions — Gliosarcoma

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group 1 (CB-NK-TGF-betaR2-/NR3C1- ) (Experimental): Participants will receive CB-NK-TGF-betaR2-/NR3C1- intratumorally over 10 minutes followed by 1 ml of Normal Saline injected over additional 10 min via Ommaya catheter every four weeks for up to 8 doses in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: Cord Blood-derived Expanded Allogeneic Natural Killer Cells
- Group 2 (CB-NK-TGF-betaR2-/NR3C1-, resection) (Experimental): Ommaya catheter will be inserted prior to the 1st injection of NK cells (at the time of screening biopsy). Two weeks prior to Surgical resection participants will receive the 1st dose of CB-NK-TGF-betaR2-/NR3C1- intratumorally over 10 minutes followed by 1 ml of Normal Saline injected over an additional 10 min via Ommaya catheter. Ommaya catheter will be taken out at the time of standard of care surgical resection of the tumor on day 15 and then another one will be inserted at the end of surgery for future IT injections. Beginning 2 weeks after surgery, participants will receive CB-NK-TGF-betaR2-/ NR3C1- intratumorally over 10 minutes followed by 1 ml of Normal Saline injected over additional 10 min via Ommaya catheter every 4 weeks for up to 7 doses (total of 8 doses) in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: Cord Blood-derived Expanded Allogeneic Natural Killer Cells; Procedure: Resection

INTERVENTIONS:
Biological: Cord Blood-derived Expanded Allogeneic Natural Killer Cells — Given CB-NK-TGF-betaR2-/NR3C1- intratumorally
  Other Names: Allogeneic CB-derived Ex vivo-expanded NK Cells; CB-derived Expanded Allogeneic NK Cells; UCB-derived Expanded Allogeneic NK Cells; Umbilical Cord Blood-derived Expanded Allogeneic Natural Killer Cells
Procedure: Resection — Undergo surgical resection
  Other Names: Surgical Resection
  Arms: Group 2 (CB-NK-TGF-betaR2-/NR3C1-, resection)

SUMMARY:
This phase I trial is to find out the best dose, possible benefits and/or side effects of engineered natural killer (NK) cells containing deleted TGF-betaR2 and NR3C1 (cord blood [CB]-NK-TGF-betaR2-/NR3C1-) in treating patients with glioblastoma that has come back (recurrent). CB-NK-TGF-betaR2-/NR3C1- cells are genetically changed immune cells that may help to control the disease.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

* To determine the safety and tolerability of intratumoral injection of escalating doses of allogeneic CB-NK-TGF-£]R2-/NR3C1- in patients with recurrent grade 4 astrocytoma,
* To determine the maximum tolerated dose (MTD) and the occurrence of dose limiting toxicities (DLTs) (Group 1) of CB-NK-TGF-£]R2-/NR3C1- administered via IT injection in patients with recurrent grade 4 astrocytoma
* To evaluate the immunological phenotype and anti-tumor function of NK cells in resected tumor tissue after treatment with CB-NK-TGF-âR2-/NR3C1- in the surgical expansion group (Group 2). Persistency of the NK cells in the tissue will be assessed by flow cytometry. Tissue cells will be stained with anti human CD45, anti human CD56 and anti HLA molecule expressed by the cord blood donor infused in the patient. NK cells from the tissue may be isolated using magnetic bead selection (anti-HLA specific from cord blood donor labeled with PE and them use a anti PE magnetics bead selection). Those NK cells would be used to perform a chromium release assay (killing assay) to test the ability of the NK in killing K562 and GSC targets. If the NK cells obtained from the tissue are too low to do killing assay, the NK cells could be expanded for one week using UAPC and IL2 to get more NK cells for assays.

SECONDARY OBJECTIVE:

-To determine response as measured by Response Assessment in Neuro-Oncology (RANO), duration of clinical response, progression free survival (PFS), time to progression (TTP), and overall survival (OS)ƒn

EXPLORATORY OBJECTIVES:

-Monitoring immune responses following CB-NK-TGF-£]R2-/NR3C1- dosing, in vivo persistence and expansion of CB-NK-TGF-£]R2-/NR3C1- during treatment, characterization of immune cell subpopulations in the peripheral blood, serum analysis of immune correlates, alloreactivity characterization, and anti-HLA antibody analysis, and CB-NK-TGF-£]R2-/NR3C1- trafficking in tumor microenvironments in the surgical expansion cohort. Tumor tissue from surgical resection will be further analyzed for immune infiltrates, fibrosis, and tumor microenvironment.

ELIGIBILITY:
Inclusion Criteria

1. Signed and dated informed consent.
2. Male or female participants aged ≥ 12 years on the day of signing informed consent.
3. Has histologically confirmed supratentorial World Health Organization grade 4 recurrent astrocytoma to include recurrent IDH WT glioblastoma or gliosarcoma and recurrent IDHmutant grade 4 astrocytoma, and recurrent gliosarcoma with any prior number of recurrences, and who have received prior radiation and temozolomide therapy. Participants will be eligible if the original histology was lower-grade glioma grade 2 or 3 and a subsequent histological diagnosis of recurrent glioblastoma or IDH-mutant grade 4 astrocytoma is made.
4. Karnofsky Performance Score (KPS) of >70 at trial entry. Lansky >70 at trial entry for patients less than 16.
5. Must be at least 12 weeks from receiving conformal radiation, unless RANO criteria for early progression are met.
6. A baseline brain MRI with Advance Brain Tumor Imaging (ABTI) must be obtained no more than 30 days prior to study registration
7. Patients having undergone recent surgery are eligible so long as they are at least 3 weeks from resection or at least 1 week from stereotactic biopsy and recovered from any operative or perioperative complications.
8. Adequate hematological function defined by white blood cell (WBC) count ≥ 3 x 10°9/L with absolute neutrophil count (ANC) ≥ 1.5 x 10°9/L, lymphocyte count ≥ 0.5 x 10°9/L, platelet count ≥ 100 x 10°/L, and Hgb ≥ 9 g/ dL (in absence of blood transfusion).
9. Adequate hepatic function defined by a total bilirubin level ≤ 1.5 x ULN, an AST level ≤ 2.5 x ULN, and an ALT level ≤ 2.5 x ULN, and INR ≤ 1.5 10. Adequate renal function defined creatinine ≥ 1.5 X upper limit of normal (ULN) OR creatinine clearance ≥ 60 mL/min for participant with creatinine levels > 1.5 X institutional ULN

11. Female participant of childbearing potential should have a negative serum pregnancy test within 14 days (+/-2 working days) of study registration.

12. Female participants of childbearing potential should be willing to use 2 methods of birth control or be surgically sterile, or abstain from heterosexual activity for the course of the study and for 3 months after the last dose of study therapy. Participants of childbearing potential are those who have not been surgically sterilized or have not been free from menses for > 1 year.

13. Male participants should agree to use 2 methods of highly effective contraception starting with the first dose of study therapy and for 3 months after the last dose of study therapy.

14. For the surgical expansion group (Group 2): there must be at least 1 cm2 of contrast-enhancing disease that is considered resectable by the neurosurgeon.

Exclusion Criteria

1. Has received prior therapy with Gliadel or bevacizumab.
2. Has received prior interstitial brachytherapy, implanted chemotherapy, or therapeutics delivered by local injection or convection enhanced delivery.
3. Is currently participating in or has participated in a study of cancer directed investigational agent or using an investigational device within 4 weeks since last dose of agent administration or device use, or is planning to continue or start treatment with Optune® during participation in this trial.
4. Has known severe hypersensitivity to monoclonal antibodies, any history of anaphylaxis, or recent, within 5 months, history of uncontrolled asthma.
5. Has a known history of Human Immunodeficiency Virus (HIV) (positive HIV 1/2 antibodies); HTLV1 and/or HTLV2; active Hepatitis B (e.g., HbsAg reactive) or Hepatitis C (e.g., HCV RNA [qualitative] is detected). Patients with prior HBV vaccination (anti-HBs positive, HbsAg negative, anti-HBc negative) will NOT be excluded.
6. Has a diagnosis of immunodeficiency or is receiving any immunosuppressive therapy within 7 days prior to study registration.
7. Has had prior chemotherapy or targeted small molecule therapy within 2 weeks prior to study Day 0.

   1. Note: Participants with ≤ Grade 2 neuropathy are an exception to this criterion and may qualify for the study.
   2. Note: If participant received major surgery (other than craniotomy), they must have recovered adequately from the toxicity and/or complications from the intervention prior to starting therapy.
8. Has had prior radiation therapy less than 12 weeks prior to study registration, unless RANO criteria for early progression are met.
9. Has had prior therapy with any antibody/drug targeting T cell co-regulatory proteins (immune checkpoints) such as anti-PD-1, anti-PD-L1, or anti-CTLA-4 antibody within the last three months prior to study registration -.
10. Has a known additional malignancy that is progressing or requires active treatment.

    Exceptions include but are not limited to basal cell carcinoma of the skin, squamous cell carcinoma of the skin, or in situ cervical cancer that has undergone potentially curative therapy. Any exceptions must be discussed with the protocol PI.
11. Has known gliomatous cerebri, extracranial disease, or tumor localized primarily to the brainstem or spinal cord.
12. Brain midline shift greater than 0.5 cm or pending herniation seen on baseline MRI ABTI.
13. Tumors larger than 5 cm at greatest diameter
14. Has an active autoimmune disease requiring systemic treatment within the past 3 months or a documented history of clinically severe autoimmune disease, or a syndrome that requires systemic steroids or immunosuppressive agents. Participants with vitiligo or resolved childhood asthma/atopy would be an exception to this rule. Participants that require intermittent use of bronchodilators or local steroid injections would not be excluded from the study. Participants with hypothyroidism stable on hormone replacement or Sjogren's syndrome will not be excluded from the study.
15. Has evidence of interstitial lung disease or active, non-infectious pneumonitis.
16. Has an active infection requiring systemic therapy or that in the opinion of the PI may interfere with the participant's participation, assessment of experimental treatment toxicity or increase the participant's risk of side effects.
17. Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the participant's participation for the full duration of the trial, or is not in the best interest of the participant to participate in the opinion of the treating investigator.
18. Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
19. Is pregnant, breastfeeding, or expecting to conceive or father children within the projected duration of the trial, starting with the screening visit and through 3 months after last dose of the study treatment.
20. Has received a live vaccine within 30 days prior to the first dose of trial treatment.
21. Has a contraindication for undergoing MRIs.
22. Has evidence of bleeding diathesis or coagulopathy.
23. Is on full dose anticoagulants or antiplatelet therapy that cannot be held.
24. Has significant hemorrhage on baseline MRI ABTI defined as >1 cm diameter of acute blood.
25. Has received any organ transplantation, including allogeneic stem-cell transplantation, but with the exception of transplants that do not require immunosuppression (e.g., corneal transplant, hair transplant).
26. Has multicentric disease. Subject has multicentric GBM, defined as discrete sites of contrast enhancing disease without contiguous T2/FLAIR abnormality that require distinct radiotherapy ports. Satellite lesions that are associated with a contiguous area of T2/FLAIR abnormality as the main lesion(s) and that are encompassed within the same radiotherapy port as the main lesion(s) are permitted.

Treatment will be up to 32 weeks in duration.

The number of cells administered will be based on gene editing efficiency. CB-NK-TGF-£]R2-/NR3C1-cells will be administered via intraventricular injection via an Ommaya reservoir on day 0 and every 4 weeks y for up to 8 doses total in Group 1.

Surgical patients in Group 2 will undergo intraventricular insertion of an Ommaya (day -14 to -

1). They will then undergo IT injection via the Ommaya reservoir of CB-NK-TGF-£]R2-/NR3C1-cells on day 0. Prior to planned tumor resection to occur between days 7-14. Every 4 week intraventricular injections of CB-NK-TGF-£]R2-/NR3C1- cells will be administered for a total of 8 intraventricular treatments.

In the setting of any surgical complications following Ommaya placement, CB-NK-TGF-£]R2-/NR3C1- cells may be delayed and administered once the patient is deemed stable by the neurosurgeon following Ommaya placement.

Treatment will continue until tumor progression or intolerable toxicity, or a maximum of 8 intraventricular treatments with CB-NK-TGF-£]R2-/NR3C1- cells whichever occurs first.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2023-04-28 (Actual); Primary Completion 2027-01-31 (Estimated); Study Completion 2027-01-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of dose-limiting toxicities (DLTs) (Group 1) | Up to 28 days
  Will determine maximum tolerated dose and safety of escalating doses of cord blood (CB)-(NK) cells patients with recurrent glioblastoma. A DLT is defined as any grade >= 3 adverse event assessed as related to CB-NK cells by the investigator (that is, grade >= 3 adverse drug reaction; grading according to the National Cancer Institute-Common Terminology Criteria for Adverse Events version 4.03.

SECONDARY OUTCOMES:
Overall survival (OS) | From definitive histological diagnosis until the time of death, assessed up to 90 days post-treatment
  OS will be estimated using the Kaplan-Meier method and the comparison between or among patients' characteristics groups will be evaluated by log-rank test. Cox regression models will be applied to assess the effect of covariates of interest on OS.
Objective response rate (ORR) | Up to 90 days post-treatment
  ORR will be defined as the proportion of patients with tumor size reduction (partial response and complete response, per Response Assessment in Neuro-Oncology [RANO] criteria). Will be calculated as the ratio of number of patients with response over number of patients treated, and 95% confidence interval of ORR will be estimated.
Duration of response (DOR) | From the time of initial response until documented tumor progression per RANO criteria, assessed up to 90 days
Time to progression (TTP) | From the date of start of treatment until the tumor progression as defined by RANO, assessed up to 90 days post-treatment
  TTP will be estimated using the Kaplan-Meier method and the comparison between or among patients' characteristics groups will be evaluated by log-rank test. Cox regression models will be applied to assess the effect of covariates of interest on TTP.
Progression-free survival (PFS) | From the start of treatment until the time of first disease progression or relapse (as defined by RANO criteria), or death due to disease, assessed up to 6 months post-treatment
  PFS will be estimated using the Kaplan-Meier method and the comparison between or among patients' characteristics groups will be evaluated by log-rank test. Cox regression models will be applied to assess the effect of covariates of interest on PFS. The point estimate of median PFS and 6-month progression-free survival (PFS6) will be estimated.

CONTACTS AND LOCATIONS:
Overall Officials: Shiao-Pei S Weathers, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center — http://www.mdanderson.org